CLINICAL TRIAL: NCT04960631
Title: Evaluation of Clinical Significance and Feasibility of CT Guided Biopsy of Double Site Lesions：A Preliminary Lung Centered Study
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2018060
Record Dates: First submitted 2021-06-29; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-06

CONDITIONS: Carcinoma of the Lungs

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clinical diagnosis of suspected malignant tumor by dual site CT guided needle biopsy
  Interventions: Diagnostic Test: Double site CT guided needle biopsy

INTERVENTIONS:
Diagnostic Test: Double site CT guided needle biopsy — Double site CT guided needle biopsy

SUMMARY:
This study aims to explore the clinical significance and feasibility of double site biopsy by analyzing the pathological characteristics and the incidence of main complications of CT guided puncture biopsy of lung and other parts coexisting lesions.

DETAILED DESCRIPTION:
CT guided biopsy is minimally invasive, accurate and low cost. It is often used as an important diagnostic method when the clinical suspect of malignant disease or the treatment effect of the disease is not good. In patients with suspected malignant lung disease, metastasis of other parts of lung, pulmonary door, mediastinum, bone, and distant soft tissue may be combined at the same time. It is the key link of clinical work to evaluate the nature of these coexisting lesions accurately and choose appropriate treatment methods. At present, there is little clinical study on lung centered double site biopsy. This study aims to explore the clinical significance and feasibility of double site biopsy by analyzing the pathological characteristics and the incidence of main complications of CT guided puncture biopsy of lung and other parts coexisting lesions.

ELIGIBILITY:
Inclusion Criteria:

* patients with suspected malignancy
* underwent dual site CT guided biopsy in the Third Hospital of Peking University

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinical data of 134 consecutive patients with suspected malignancy who underwent dual site CT guided biopsy in the Third Hospital of Peking University from January 2011 to October 2014
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
for the combination of two site biopsies | up to 2weeks
  The incidence of 4 kinds of combined pathological results in different lesion location groups was analyzed.
for the combination of two site biopsy approaches 1 | up to 2weeks
  The incidence of pneumothorax on the surgical side after unilateral lung biopsy
for the combination of two site biopsy approaches 2 | up to 2weeks
  the incidence of pneumothorax on the surgical side after bilateral lung biopsy
for the combination of two site biopsy approaches 3 | up to 2weeks
  the incidence of intra tissue hemorrhage after biopsy were statistically analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Huishu Huishu, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No